CLINICAL TRIAL: NCT02119676
Title: A Randomized, Double-Blind Study of Ruxolitinib or Placebo in Combination With Regorafenib in Subjects With Relapsed or Refractory Metastatic Colorectal Cancer
Brief Title: Study of Ruxolitinib in Colorectal Cancer Patients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Substudy 1 was terminated for futility at interim analysis and Substudy 2 was terminated per sponsor decision.
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB18424-267
Record Dates: First submitted 2014-04-17; First posted 2014-04-22 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2018-02-13 (Actual); Status verified 2018-01

CONDITIONS: CRC (Colorectal Cancer)
Keywords: Metastatic Colorectal Cancer; Colon Cancer; Ruxolitinib; adenocarcinoma; regorafenib; Jakavi ®; Jakafi ®; Stivarga ®
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Adenocarcinoma | interventions — ruxolitinib; regorafenib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ruxolitinib plus regorafenib (Experimental)
  Interventions: Drug: Ruxolitinib; Drug: Regorafenib
- Placebo plus regorafenib (Active Comparator)
  Interventions: Drug: Regorafenib; Drug: Placebo

INTERVENTIONS:
Drug: Ruxolitinib — 5 mg tablets to be administered by mouth
  Ruxolitinib 20 mg twice a day (BID) (Part 1) (NOTE: The starting dose for the randomized portion of study (Part 2) was 15 mg BID based on results from Part 1.)
  Other Names: Jakafi ®; Jakavi ®
  Arms: Ruxolitinib plus regorafenib
Drug: Regorafenib — Regorafenib 160mg once daily for the first 21 days of each 28-day cycle. (NOTE: Dose interruptions and modifications for regorafenib are expected when toxicities occur in which dose interruptions or modifications are appropriate.)
  Other Names: Stivarga ®
Drug: Placebo — 5 mg matching placebo tablets to be administered by mouth
  Arms: Placebo plus regorafenib

SUMMARY:
The purpose of this study was to determine if ruxolitinib, in combination with regorafenib, is safe and effective in the treatment of metastatic colorectal cancer.

DETAILED DESCRIPTION:
The study consisted of an open-label, Part 1 safety run-in (consisting of 1 to 3 cohorts of 9 subjects each), to confirm the safety of the regorafenib/ruxolitinib combination in subjects with relapsed or refractory metastatic colorectal cancer (CRC). If determined to be tolerable, Part 2 was to proceed as a randomized, double-blind study evaluating ruxolitinib or placebo in combination with regorafenib in subjects with relapsed or refractory metastatic CRC previously treated with fluoropyrimidine, oxaliplatin, and/or irinotecan based chemotherapy, an anti-vascular endothelial growth factor (VEGF) therapy and if Kirsten rat sarcoma (KRAS) wild type an anti-epidermal growth factor receptor (EGFR) therapy.

Subjects in the safety run-in received open-label ruxolitinib and regorafenib; for the randomized, double-blind portion of the study all subjects received regorafenib and either ruxolitinib or placebo in a 1:1 blinded manner. Treatment for all subjects consisted of repeating 28-day cycles. Regorafenib was self-administered for the first 21 days of each cycle, and ruxolitinib/placebo was self-administered during the entire 28-day cycle. Treatment cycles continued as long as the regimen is tolerated, and the subject does not meet the discontinuation criteria. When subjects discontinued regorafenib, ruxolitinib or placebo they remained in the study and were followed for subsequent treatment regimens which were initiated and survival.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed adenocarcinoma of the colon or rectum that is metastatic.
* Previous treatment with fluoropyrimidine-, oxaliplatin- and irinotecan- based chemotherapy, an anti-VEGF therapy (if no contraindication) and if KRAS wild type and no contraindication, an anti-EGFR therapy.
* Radiographically measurable or evaluable disease (per RECIST v1.1)
* Life expectancy of ≥ 12 weeks.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
* Three or more weeks have elapsed from the completion of previous treatment regimen and subjects must have recovered or be at a new stable baseline from any related toxicities.
* Prior radiotherapy to disease sites is allowed with certain protocol-defined restrictions.

Exclusion Criteria:

* Prior treatment with regorafenib.
* Presence of active gastrointestinal disease or other condition that will interfere significantly with the absorption of drugs.
* Active peptic ulcer disease, inflammatory bowel disease (eg, ulcerative colitis, Crohn's disease), diverticulitis, or other gastrointestinal conditions with increased risk of perforation or gastrointestinal bleeding.
* Recent history (≤ 3 months) or ongoing partial or complete bowel obstruction unless due to disease under study and corrected with surgery.
* Blood pressure ≥ 140/90 mmHg.
* Active bleeding diathesis or history of any major bleeding (eg, requiring transfusion of red blood cells (RBCs), central nervous system (CNS) bleeding, or significant hemoptysis within 6 months of enrollment. Subjects with bleeding secondary to underlying disease (including gastrointestinal (GI) perforation or fistula) that has been corrected by surgery or alternative procedure may be included.
* Clinically significant cardiac disease including unstable angina, acute myocardial infarction within 6 months from Day 1 of study drug administration, New York Heart Association Class II, III, or IV congestive heart failure, and arrhythmia requiring therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 396 (Actual)
Dates: Start 2014-03; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Albert Assad, Study Director — Incyte Corporation
Locations (86):
- United States (57):
  - Chandler, Arizona
  - Gilbert, Arizona
  - Mesa, Arizona
  - Scottsdale, Arizona
  - Los Angeles, California
  - Pasadena, California
  - Santa Barbara, California
  - Aurora, Colorado
  - Colorado Springs, Colorado
  - Denver, Colorado
  - Altamonte Springs, Florida
  - Miami, Florida
  - Ocala, Florida
  - Orlando, Florida
  - Tampa, Florida
  - Niles, Illinois
  - Lafayette, Indiana
  - Ames, Iowa
  - New Orleans, Louisiana
  - Baltimore, Maryland
  - Jefferson City, Missouri
  - St Louis, Missouri
  - Lincoln, Nebraska
  - Omaha, Nebraska
  - Henderson, Nevada
  - Las Vegas, Nevada
  - Albany, New York
  - Binghamton, New York
  - Hudson, New York
  - Johnson City, New York
  - New York, New York
  - The Bronx, New York
  - Canton, Ohio
  - Cincinnati, Ohio
  - Portland, Oregon
  - Charleston, South Carolina
  - Easley, South Carolina
  - Greenville, South Carolina
  - Greer, South Carolina
  - Sumter, South Carolina
  - Chattanooga, Tennessee
  - Nashville, Tennessee
  - Arlington, Texas
  - El Paso, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - Paris, Texas
  - Plano, Texas
  - Tyler, Texas
  - American Fork, Utah
  - Bountiful, Utah
  - Murray, Utah
  - Provo, Utah
  - Salt Lake City, Utah
  - West Jordan, Utah
  - Roanoke, Virginia
  - Vancouver, Washington
- Australia (5):
  - Bentleigh East
  - Herston
  - Kurralta Park
  - New Lambton Heights
  - Randwick
- France (6):
  - Avignon
  - Besançon
  - Le Mans
  - Lille
  - Marseille
  - Paris
- Germany (3):
  - Augsburg
  - Halle
  - Hamburg
- Israel (5):
  - Beersheba
  - Haifa
  - Petah Tikva
  - Ramat Gan
  - Tel Aviv
- Soeul, South Korea
- Spain (5):
  - Oviedo, Principality of Asturias
  - Barcelona
  - Madrid
  - Seville
  - Valencia
- United Kingdom (4):
  - Birmingham
  - Bournemouth
  - London
  - Sutton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In Substudy 1, the first subject was enrolled on 29 OCT 2014, and the last subject was enrolled on 23 JUL 2015. In Substudy 2, the first subject was enrolled on 05 NOV 2014, and the last subject was enrolled on 02 OCT 2015.
Pre-assignment Details: Substudy 1; 4 participants were assigned a randomization number but were not given study drug because of clinical deterioration or withdrawal of consent. Substudy 2; 9 participants were assigned a randomization number, but weren't given study drug due to clinical deterioration, withdrawal of consent or not meeting all of the eligibility criteria.
Groups:
- Substudy 1: Ruxolitinib + Regorafenib: Ruxolitinib 15 mg twice a day (BID) continuous with regorafenib 160 mg once daily (QD) for the first 21 days of each 28-day cycle.
- Substudy 1: Placebo + Regorafenib; Substudy 2: Placebo + Regorafenib: Placebo BID continuous with regorafenib 160 mg QD for the first 21 days of each 28-day cycle.
- Substudy 2: Ruxolitinib + Regorafenib: Ruxolitinib 15 mg BID continuous with regorafenib 160 mg QD for the first 21 days of each 28-day cycle.
Period: Overall Study
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Started | 87 | 88 | 110 | 111
Treated Patients | 85 | 86 | 106 | 106
Completed (Ongoing treatment at time of termination. Termination=Substudy 1: 27Jan2016; Substudy 2: 11Feb2016.) | 4 | 2 | 13 | 10
Not Completed | 83 | 86 | 97 | 101
Not completed — Adverse Event | 9 | 17 | 10 | 10
Not completed — Disease progression | 53 | 55 | 68 | 73
Not completed — Patient decision, inc. consent withdrawn | 4 | 5 | 5 | 6
Not completed — Physician Decision | 4 | 2 | 3 | 2
Not completed — Death | 9 | 3 | 2 | 1
Not completed — Noncompliance | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Protocol deviation | 0 | 0 | 1 | 0
Not completed — Other, unspecified | 2 | 1 | 3 | 4
Not completed — Did not receive study med | 2 | 2 | 4 | 5

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population consisted of participants that were randomized in the study.
Groups:
- Substudy 1: Ruxolitinib + Regorafenib; Substudy 2: Ruxolitinib + Regorafenib: Ruxolitinib 15 mg BID continuous with regorafenib 160 mg QD for the first 21 days of each 28-day cycle.
- Total: Total of all reporting groups
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib | Total
Number analyzed (Participants) | 87 | 88 | 110 | 111 | 396
Age, Continuous [Mean (Full Range); unit: years] | 60.8 [34.0 to 84.0] | 59.5 [36.0 to 81.0] | 59.0 [37.0 to 79.0] | 59.2 [19.0 to 83.0] | 59.6 [19 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 32 | 48 | 54 | 168
  Male | 53 | 56 | 62 | 57 | 228
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 10 | 9 | 21
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 0 | 1
  Black or African American | 7 | 7 | 6 | 7 | 27
  White | 70 | 70 | 84 | 80 | 304
  More than one race | 10 | 9 | 5 | 11 | 35
  Unknown or Not Reported | 0 | 0 | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from randomization to death due to any cause. Participants without death observed at the time of the analysis will be censored at last date known to be alive. The median overall survival time was estimated using the Kaplan-Meier method. Overall survival was compared between treatment groups using log-rank test.
Time Frame: Baseline until death due to any cause; up to 16 months or data cut-off 11 FEB 2016.
Population: Intent-to-treat (ITT) population included all subjects randomized in Substudy 1 and Substudy 2 of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 87 | 88 | 110 | 111
months | 4.6 [3.5 to 5.4] | 5.3 [4.3 to 6.0] | 11.4 [9.0 to 13.2] | 10.9 [7.2 to NA] — Not estimable due to insufficient number of participants with events.
Statistical Analysis 1: Comparison: Substudy 1: Ruxolitinib + Regorafenib vs Substudy 1: Placebo + Regorafenib; Test type: Other; p = 0.588, Log Rank — 1-sided; Log-rank test stratified by modified Glasgow Prognostic Score (mGPS) and geographical region; Hazard Ratio (HR) = 1.04, 95% CI 2-sided [0.73 to 1.49] — Estimated using a Cox regression model with Efron's method used for ties, stratified by mGPS score and geographical region
Statistical Analysis 2: Comparison: Substudy 2: Ruxolitinib + Regorafenib vs Substudy 2: Placebo + Regorafenib; Test type: Other; p = 0.136, Log Rank — 1-sided; Log rank test stratified by geographical region; Hazard Ratio (HR) = 0.77, 95% CI 2-sided [0.48 to 1.23] — Estimated using Cox regression model with Efron's method used for ties, stratified by geographical region

2. Secondary Outcome: Progression Free Survival (PFS)
Description: Progressive Disease (PD) is defined using Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 at least a 20% increase in the sum of the Longest Diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions, unequivocal progression of non-target lesions, or the appearance of new lesions.
Time Frame: Baseline through disease progression, or death due to any cause if sooner; up to 16 months or data cut-off 11 FEB 2016.
Population: Intent-to-treat (ITT) population included all subjects randomized in Substudy 1 and Substudy 2 of the study.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 87 | 88 | 110 | 111
months | 2.2 [1.9 to 3.0] | 2.1 [1.8 to 2.7] | 3.5 [3.0 to 3.8] | 2.0 [1.9 to 3.1]

3. Secondary Outcome: Overall Response Rate (ORR)
Description: Response defined per Response Evaluation Criteria In Solid Tumors (RECIST) criteria: Complete Response (CR)=disappearance of all target and non-target lesions without new lesion; Partial Response (PR)=30% decrease in sum of longest diameter of target lesions, non-target lesion not progressed, and no new lesion; Progressive Disease=20% increase in sum of longest diameter of target lesions, or non-target lesion progression, or identification of new lesion; Stable Disease=small changes that do not meet above criteria. ORR was defined as the proportion of participants who achieved a best response of either CR or PR. ORR=number of participants with CR or PR/number of participants randomized.
Time Frame: Baseline through end of study; up to 16 months or data cut-off 11 FEB 2016.
Population: Intent-to-treat (ITT) population included all subjects randomized in Substudy 1 and Substudy 2 of the study.
Measure: Number (95% Confidence Interval); unit: percentage of responders
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 87 | 88 | 110 | 111
percentage of responders | 0.0 [0.0 to 4.2] | 0.0 [0.0 to 4.1] | 2.7 [0.6 to 7.8] | 4.5 [1.5 to 10.2]

4. Secondary Outcome: Duration of Response
Description: Duration of response is defined as the time from response (CR/PR) until the earliest date of disease progression determined by investigator assessment of objective radiographic disease assessments per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death due to any cause.
Time Frame: Baseline through end of study; up to 16 months or data cut-off 11 FEB 2016.
Population: No data displayed because outcome measure has not been analyzed. Duration of response analyses was not done since there were no responders in Substudy 1 and very few responders in Substudy 2 at data cutoff (27JAN2016 for Substudy 1 and 11Feb2016 for Substudy 2). Duration of response analysis was not done in both substudies.
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 0 | 0 | 0 | 0

5. Secondary Outcome: Percentage of Participants Achieving Disease Control
Description: Disease control as measured by the percentage of participants whose best response was complete response (CR), partial response (PR), or stable disease (SD) per RECIST v.1.1.
Time Frame: Baseline through end of study; up to 16 months or data cut-off 11 FEB 2016.
Population: Intent-to-treat (ITT) population included all subjects randomized in Substudy 1 and Substudy 2 of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 87 | 88 | 110 | 111
percentage of participants | 40.2 [29.9 to 51.3] | 34.1 [24.3 to 45.0] | 61.8 [52.1 to 70.9] | 36.9 [28.0 to 46.6]

6. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: TEAEs were defined as any adverse event (AE) during the study that began or worsened on or after the date of first dose of investigational product.
Time Frame: Baseline through approximately 30 days post treatment discontinuation;up to 16 months or data cut-off 27JAN 2016 for Substudy 1 and up to the data cut-off of 11FEB2016 for Substudy 2.
Population: Safety Population consists of all enrolled participants that received at least one dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Number analyzed (Participants) | 85 | 86 | 106 | 106
percentage of participants
  Participants with any TEAEs | 100.0 | 100.0 | 100.0 | 99.1
  Participants with Grade 3/4 TEAEs | 82.4 | 81.4 | 77.4 | 72.6
  Participants with any serious TEAE | 57.6 | 48.8 | 34.9 | 34.9
  Participants with a fatal TEAE | 15.3 | 9.3 | 1.9 | 3.8
  Participants who discontinued drug due to of TEAEs | 14.1 | 19.8 | 11.3 | 10.4

ADVERSE EVENTS:
Time Frame: From the first dose of study medication up to 16 months or data cut-off 11 FEB 2016.
Description: The safety evaluable population consisted of all participants exposed to at least 1 dose of study drug.
Arm/Group | Substudy 1: Ruxolitinib + Regorafenib | Substudy 1: Placebo + Regorafenib | Substudy 2: Ruxolitinib + Regorafenib | Substudy 2: Placebo + Regorafenib
Serious Adverse Events (participants affected / at risk) | 49/85 | 42/86 | 37/106 | 37/106
Other Adverse Events (participants affected / at risk) | 85/85 | 86/86 | 106/106 | 105/106
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1: Ruxolitinib + Regorafenib (N=85) | Substudy 1: Placebo + Regorafenib (N=86) | Substudy 2: Ruxolitinib + Regorafenib (N=106) | Substudy 2: Placebo + Regorafenib (N=106)
Hyperthyroidism (Endocrine disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 6 | 7 | 4 | 5
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Bloody peritoneal effluent (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematemesis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 2 | 1 | 2
Intestinal perforation (Gastrointestinal disorders) | 2 | 0 | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 2 | 1 | 3
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 1 | 0 | 5
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Subileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 4 | 3 | 4
Asthenia (General disorders) | 2 | 1 | 1 | 0
Disease progression (General disorders) | 2 | 0 | 0 | 0
General physical health deterioration (General disorders) | 4 | 3 | 1 | 1
Malaise (General disorders) | 0 | 1 | 0 | 0
Multi-organ failure (General disorders) | 0 | 1 | 0 | 0
Obstruction (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Pain (General disorders) | 0 | 3 | 1 | 1
Pyrexia (General disorders) | 3 | 2 | 1 | 3
Systemic inflammatory response syndrome (General disorders) | 1 | 0 | 1 | 0
Hepatobiliary disorders (General disorders) | 5 | 2 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0 | 0 | 0
Hepatorenal syndrome (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 2 | 1 | 0 | 1
Arthritis infective (Infections and infestations) | 0 | 1 | 0 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Biliary sepsis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0 | 0
Hepatic infection bacterial (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 2 | 1 | 0 | 0
Liver abscess (Infections and infestations) | 1 | 0 | 0 | 0
Perirectal abscess (Infections and infestations) | 1 | 0 | 0 | 0
Peritonitis (Infections and infestations) | 0 | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 5 | 2 | 0 | 0
Sepsis (Infections and infestations) | 6 | 1 | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 1 | 2 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 4 | 1 | 0 | 3
Blood creatinine increased (Investigations) | 1 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Hepatic enzyme abnormal (Investigations) | 0 | 1 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 1 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 3 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrospinal fistula (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 1 | 1 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Lacunar infarction (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0 | 0
Completed suicide (Psychiatric disorders) | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 1 | 0 | 0
Vesical fistula (Renal and urinary disorders) | 0 | 1 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 5 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Embolism venous (Vascular disorders) | 0 | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 2 | 2 | 0
Hypotension (Vascular disorders) | 1 | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 2 | 0
Biliary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Endocarditis (Infections and infestations) | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Platelet count decreased (Investigations) | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Spinal cord compression (Nervous system disorders) | 0 | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 1
VIIth nerve paralysis (Nervous system disorders) | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Renal injury (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal vein thrombosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 1
Lower respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Embolism (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Substudy 1: Ruxolitinib + Regorafenib (N=85) | Substudy 1: Placebo + Regorafenib (N=86) | Substudy 2: Ruxolitinib + Regorafenib (N=106) | Substudy 2: Placebo + Regorafenib (N=106)
Anaemia (Blood and lymphatic system disorders) | 10 | 12 | 27 | 12
Hypothyroidism (Endocrine disorders) | 2 | 6 | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 21 | 24 | 24 | 26
Abdominal pain upper (Gastrointestinal disorders) | 4 | 6 | 6 | 11
Ascites (Gastrointestinal disorders) | 6 | 2 | 2 | 7
Constipation (Gastrointestinal disorders) | 27 | 21 | 24 | 22
Diarrhoea (Gastrointestinal disorders) | 32 | 27 | 41 | 29
Dry mouth (Gastrointestinal disorders) | 3 | 6 | 4 | 4
Flatulence (Gastrointestinal disorders) | 5 | 6 | 5 | 5
Nausea (Gastrointestinal disorders) | 22 | 22 | 30 | 22
Stomatitis (Gastrointestinal disorders) | 21 | 18 | 19 | 21
Vomiting (Gastrointestinal disorders) | 16 | 20 | 24 | 15
Asthenia (General disorders) | 22 | 22 | 19 | 23
Chills (General disorders) | 2 | 5 | 5 | 4
Fatigue (General disorders) | 29 | 31 | 43 | 47
Oedema peripheral (General disorders) | 8 | 9 | 2 | 8
Pain (General disorders) | 5 | 4 | 3 | 6
Pyrexia (General disorders) | 16 | 15 | 20 | 16
Hyperbilirubinaemia (Hepatobiliary disorders) | 5 | 3 | 4 | 5
Urinary tract infection (Infections and infestations) | 11 | 6 | 8 | 8
Alanine aminotransferase increased (Investigations) | 5 | 8 | 8 | 11
Aspartate aminotransferase increased (Investigations) | 8 | 14 | 12 | 13
Blood alkaline phosphatase increased (Investigations) | 4 | 6 | 4 | 5
Blood bilirubin increased (Investigations) | 12 | 12 | 7 | 15
Lipase increased (Investigations) | 1 | 5 | 5 | 5
Weight decreased (Investigations) | 13 | 15 | 13 | 16
Decreased appetite (Metabolism and nutrition disorders) | 31 | 31 | 28 | 35
Dehydration (Metabolism and nutrition disorders) | 11 | 7 | 8 | 12
Hypoalbuminaemia (Metabolism and nutrition disorders) | 3 | 6 | 1 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 6 | 6 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 11 | 5 | 8 | 13
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 5 | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 15 | 11 | 14 | 11
Muscle spasms (Musculoskeletal and connective tissue disorders) | 7 | 2 | 9 | 11
Muscular weakness (Musculoskeletal and connective tissue disorders) | 5 | 0 | 3 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 5 | 7 | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 2 | 10 | 10
Dizziness (Nervous system disorders) | 4 | 5 | 11 | 5
Dysgeusia (Nervous system disorders) | 6 | 6 | 6 | 4
Headache (Nervous system disorders) | 13 | 16 | 21 | 26
Insomnia (Psychiatric disorders) | 7 | 5 | 11 | 5
Pollakiuria (Renal and urinary disorders) | 6 | 1 | 2 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 8 | 10 | 7
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 11 | 14 | 22 | 27
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 14 | 15 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 6 | 4 | 4 | 10
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 5 | 7 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 6 | 3 | 3
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 6 | 8 | 10
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 36 | 38 | 61 | 50
Pruritus (Skin and subcutaneous tissue disorders) | 5 | 3 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 8 | 12 | 15 | 12
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 5 | 2 | 5
Hypertension (Vascular disorders) | 18 | 22 | 44 | 42
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 1 | 4 | 6
Abdominal distension (Gastrointestinal disorders) | 2 | 4 | 1 | 7
Chest pain (General disorders) | 3 | 3 | 7 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4 | 3 | 6 | 5
Neuropathy peripheral (Nervous system disorders) | 2 | 2 | 9 | 6

LIMITATIONS AND CAVEATS:
Substudy 1 was terminated for futility at interim analysis and Substudy 2 was terminated per sponsor decision.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.